CLINICAL TRIAL: NCT01520259
Title: A Pilot Study of Gallbladder Cancer in Chile
Brief Title: Initial Study of Gallbladder Cancer in Chile
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912020; 12-C-N020
Record Dates: First submitted 2012-01-26; First posted 2012-01-27 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2019-08-08

CONDITIONS: Gallbaldder Cancer
Keywords: Gallbaldder; Gallstones; Inflammation; Cholecystectomy; Cancer; Gallbaldder Cancer
MeSH Terms: conditions — Gallstones; Inflammation; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cases: Women from the cohort with gallbladder cancer
- cohort: Women from Chile screened for gallbladder cancer with and without gallstones
- controls: Women from the cohort with gallstones

SUMMARY:
Background:

- Chile has the highest diagnosis and death rates of gallbladder cancer in the world. Gallbladder cancer is also the leading cause of cancer death in Chilean women. High rates of gallstones and obesity, as well as genetic concerns, may explain these high rates. Researchers want to study gallbladder cancer in more depth in Chile. A small study must be done to see if a full-scale study is feasible.

Objectives:

- To test the methods and procedures of a small-scale study of gallbladder cancer in Chile.

Eligibility:

* Individuals at least 18 years of age who have gallbladder cancer or gallstones, or are healthy control volunteers.
* Participants will be recruited from four clinical centers in Chile.

Design:

* Participants will be screened with a physical exam and medical history. Because gallbladder cancer has a high fatality rate, family members may be asked to provide additional medical history information if study participants die or become too ill to provide this information.
* Participants will provide blood, urine, stool, hair, fingernail, and saliva samples.
* Gallstones, bile, and tissue samples will be collected from those who have gallbladder removal surgery. Normal and tumor tissue samples will be collected as needed.
* Treatment will not be provided as part of this protocol. This is a data collection study only.

DETAILED DESCRIPTION:
Gallbladder cancer is a leading cause of cancer death among women in Chile, which has among the highest reported gallbladder cancer incidence and mortality rates in the world. Gallbladder cancer provides a particularly good model for understanding the role of inflammation in carcinogenesis since the major risk factor, gallstones, causes substantial inflammation in the gallbladder. Chile also has a high prevalence of obesity, diabetes, and metabolic syndrome, which are increasingly understood as inflammatory disorders, but the extent to which their carcinogenic effects are mediated through inflammatory pathways is unknown.

While the vast majority of gallbladder cancer cases have gallstones, only a small fraction of

gallstone patients ever develop gallbladder cancer. Since there is no way to identify this small

proportion at risk, gallstone cases are cholecystectomized, which, given large absolute numbers of individuals with gallstones, results in overtreatment of some and under-treatment of others in a high-risk area like Chile. While cholecystectomy is standard treatment for symptomatic relief, there are more people who need surgery than there are surgeons to perform them, and individuals aged 34-49 are prioritized for treatment, regardless of symptoms. This practice may lead to overtreatment among 34-49-year-olds and under treatment of individuals aged 50 and above since they have to wait longer for surgery. At the same time, about 30% of patients with a biliary colic attack will never have another attack, and cholecystectomy does not always lead to the cessation of symptoms. In addition, cholecystectomy has been associated with an increased risk of other digestive diseases. Thus, cholecystectomy may not be needed in all gallstone patients and may in fact increase the risk of cancer in some. Better predictors of risk are clearly needed.

As with other cancers, dysplasia is an important epidemiologic endpoint as the immediate precursor to cancer since the vast majority of gallbladder cancers develop through a histologic continuum of chronic cholecystitis, pseudopyloric metaplasia, incomplete intestinal metaplasia, dysplasia, and cancer. Thus, our aim is to identify risk factors for gallbladder dysplasia and cancer (GDC) and potential non-invasive risk stratification methods, such as ultrasound characteristics alone or in combination with inflammatory markers and patient characteristics, to better understand the etiology and natural history of GDC and to help inform strategies for GDC prevention.

Together with collaborators at Pontifica Universidad Catolica (PUC), we successfully completed a pilot study in Chile that was previously reviewed and approved by SAG and provided baseline data for the proposed study. Our pilot demonstrated high recruitment rates in the target enrollment area (80%) and high rates of questionnaire completion (100%), blood collection (78% population-based controls), and participant retention (93% of eligible completed a follow-up visit). Information from the pilot was used to optimize procedures for the longitudinal study. We also found that both gallstones and gallbladder cancer were associated with systemic immune alterations, which as we previously demonstrated, reflect inflammatory changes in the gallbladder detectable in bile. The next step is to demonstrate that these markers precedeGDC by longitudinally measuring their levels among gallstone patients.

We propose to prospectively assess risk factors and early detection markers for GDC by conducting the Chile Biliary Longitudinal Study (BiLS), a cohort study of 6250 individuals with gallstones from the high- risk southern-central region of Chile. Because women are twice as likely to have gallstones and twice as likely to have gallbladder cancer as men, we plan to maximize our screening efficiency and number of outcomes by screening and enrolling women only. Since Chile is conducting a general population cohort in a small town in the high-risk area, will we benefit from the infrastructure that is already in place and be able to compare the women in our study to a set of men with gallstones enrolled by the Chilean study. We plan to enroll women with gallstones over 2 years and follow them for 6 years, conducting visits every other year to collect data on the primary exposures of interest, inflammatory markers and ultrasound characteristics, as well as additional exposures of interest, such as infections, genetics, and environmental exposures (e.g., aflatoxin, pesticides). The cohort will be complemented by an incident case-control study of 300 women with gallbladder cancer and 600 controls with and without gallstones obtained from the cohort participants.

ELIGIBILITY:
-General Case Eligibility Criteria:

18 or older

no prior cancer diagnosis (except non-melanoma skin cancer)

has gallstones/gallstone disease (including cancer)

able to participate alone or have a proxy (a close family member) answer questions about him/her

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target neighborhoods in Chile in the study areas.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2012-01-10

PRIMARY OUTCOMES:
gallbladder cancer/pre-cancer | ongoing
  gallbladder cancer/pre-cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jill E. Koshiol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- Chile (4):
  - Hospital Regional de Antofagasta, Antofagasta
  - Hospital Regional De Concepcion, Concepción
  - Hospital Sorero del Rio, Santiago
  - Hospital Regional de Temuco, Temuco